CLINICAL TRIAL: NCT06573281
Title: A Phase 1, First-Time-in-Human (FTiH), Observer-blind, Randomized, Controlled Study to Evaluate the Safety, Reactogenicity and Immune Response of Various Doses of an mRNA-based Respiratory Syncytial Virus (RSV) Investigational Vaccine in Healthy Participants 18-45 Years of Age
Brief Title: A Study on the Safety and Immune Response to an mRNA-based RSV Investigational Vaccine in Healthy Adults Aged 18-45 Years
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 222261; 2024-512846-41 (EudraCT Number)
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus (RSV); RSV mRNA vaccine; Safety; Immunogenicity; Reactogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- RSV_Group A (Experimental)
  Interventions: Biological: Investigational RSV vaccine 1
- RSV_Group B (Experimental)
  Interventions: Biological: Investigational RSV vaccine 2
- RSV_Group C (Experimental)
  Interventions: Biological: Investigational RSV vaccine 3
- RSV_Group D (Experimental)
  Interventions: Biological: Investigational RSV vaccine 4
- RSV_Group E (Experimental)
  Interventions: Biological: Investigational RSV vaccine 5
- RSV_Group F (Experimental)
  Interventions: Biological: Investigational RSV vaccine 6; Drug: Placebo
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Investigational RSV vaccine 1 — Investigational RSV vaccine 1 administered intramuscularly on Day 1 and Day 30.
  Arms: RSV_Group A
Biological: Investigational RSV vaccine 2 — Investigational RSV vaccine 2 administered intramuscularly on Day 1 and Day 30.
  Arms: RSV_Group B
Biological: Investigational RSV vaccine 3 — Investigational RSV vaccine 3 administered intramuscularly on Day 1 and Day 30.
  Arms: RSV_Group C
Biological: Investigational RSV vaccine 4 — Investigational RSV vaccine 4 administered intramuscularly on Day 1 and Day 30.
  Arms: RSV_Group D
Biological: Investigational RSV vaccine 5 — Investigational RSV vaccine 5 administered intramuscularly on Day 1 and Day 30.
  Arms: RSV_Group E
Biological: Investigational RSV vaccine 6 — Investigational RSV vaccine 6 administered intramuscularly on Day 1.
  Arms: RSV_Group F
Drug: Placebo — Placebo administered intramuscularly on Day 1 and Day 30 and for RSV_Group F placebo administered only on Day 30.
  Arms: Placebo Group; RSV_Group F

SUMMARY:
The purpose of this study is to assess the reactogenicity, safety and immune response of various formulations of the RSV mRNA investigational vaccine administered in healthy participants 18-45 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary, return for follow-up visits).
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history, clinical examination and laboratory assessment at screening.
* Male or female between and including 18 and 45 years of age at the time of enrollment into the study.
* Body mass index more than or equal to (>=) 18 kg/m^2 and less than (<) 40 kg/m^2.
* Female participants of non-childbearing potential may be enrolled in the study.
* Female participants of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration period, and
  * has a negative pregnancy test (on urine sample) on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for at least 1 month after completion of the study intervention administration series.

Exclusion Criteria:

Medical conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Hypersensitivity to latex.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality.
* Recurrent history or uncontrolled neurological disorders or seizures.
* Documented HIV, HBV, or HCV-positive participant.
* Lymphoproliferative disorder or malignancy within 5 years before the first dose of study intervention administration.
* History of or current suspicion of myocarditis or pericarditis.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine, or invasive medical device) other than the study intervention during the period beginning 30 days before the first dose of study intervention administration (Day -29 to Day 1), or their planned use during the study period.
* Has previously received an investigational or approved vaccine or antibody for prevention of RSV infection.
* Planned administration/administration of a vaccine in the period starting 30 days before the first dose and ending 30 days after the last dose of study intervention administration, except for inactivated vaccines for influenza if they are received at least 14 days before the first dose or 14 days after the last study intervention administration.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other exclusion criteria

* Pregnant or lactating female participant.
* Female participant planning to become pregnant or planning to discontinue contraceptive precautions within 1 month following the last study intervention administration.
* Alcoholism or substance use disorder within the past 24 months.
* Any study personnel or their immediate dependents, family, or household members.
* Participants with extensive body markings or conditions in the deltoid region that may preclude accurate assessment of local reactogenicity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting solicited administration site events within 7 days post-Dose 1 | From Day 1 to Day 7
Number of participants reporting solicited administration site events within 7 days post-Dose 2 | From Day 30 to Day 36
Number of participants reporting solicited systemic events within 7 days post-Dose 1 | From Day 1 to Day 7
Number of participants reporting solicited systemic events within 7 days post-Dose 2 | From Day 30 to Day 36
Number of participants reporting unsolicited adverse events (AEs) within 29 days post-Dose 1 | From Day 1 to Day 29
Number of participants reporting unsolicited AEs within 29 days post-Dose 2 | From Day 30 to Day 58
Number of participants reporting serious adverse events (SAEs) | From Day 1 (Dose 1) up to Month 7 (6 months post-Dose 2)
Number of participants reporting medically attended adverse events (MAAEs) | From Day 1 (Dose 1) up to Month 7 (6 months post-Dose 2)
Number of participants reporting adverse event of special interest (AESI) | From Day 1 (Dose 1) up to Month 7 (6 months post-Dose 2)
Number of participants reporting fatal SAEs | From Day 1 (Dose 1) up to Month 13 (study end)
Number of participants reporting related SAEs | From Day 1 (Dose 1) up to Month 13 (study end)
Number of participants reporting related AESIs | From Day 1 (Dose 1) up to Month 13 (study end)
Number of participants with clinically significant hematological and biochemical abnormalities at pre-Dose 1 | At Day 1
Number of participants with clinically significant hematological and biochemical abnormalities post-Dose 1 | At Day 8
Number of participants with clinically significant hematological and biochemical abnormalities post-Dose 1 | At Day 30
Number of participants with clinically significant hematological and biochemical abnormalities post-Dose 2 | At Day 37

SECONDARY OUTCOMES:
RSV- A neutralizing titers expressed as Geometric mean titers (GMTs) | At Day 1 (pre-Dose 1), Day 8 and Day 30 (post-Dose 1), Day 37, Day 59, Month 7 and Month 13 (post-Dose 2)
RSV- B neutralizing titers expressed as GMTs | At Day 1 (pre-Dose 1), Day 8 and Day 30 (post-Dose 1), Day 37, Day 59, Month 7 and Month 13 (post-Dose 2)
Geometric mean fold increase in serum neutralizing titers against RSV-A from baseline | Day 8 and Day 30 (post-Dose 1), Day 37, Day 59, Month 7 and Month 13 (post-Dose 2) compared with baseline (Day 1, pre-Dose 1)
Geometric mean fold increase in serum neutralizing titers against RSV-B from baseline | Day 8 and Day 30 (post-Dose 1), Day 37, Day 59, Month 7 and Month 13 (post-Dose 2) compared with baseline (Day 1, pre-Dose 1)
Number of participants with seroresponse in terms of neutralizing titer against RSV-A | Day 8 and Day 30 (post-Dose 1), Day 37, Day 59, Month 7 and Month 13 (post-Dose 2) compared with baseline (Day 1, pre-Dose 1)
  Seroresponse is defined as at least a 4-fold increase compared to pre-dosing titer.
Number of participants with seroresponse in terms of neutralizing titer against RSV-B | Day 8 and Day 30 (post-Dose 1), Day 37, Day 59, Month 7 and Month 13 (post-Dose 2) compared with baseline (Day 1, pre-Dose 1)
  Seroresponse is defined as at least a 4-fold increase compared to pre-dosing titer.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Rochester, New York
- GSK Investigational Site, Camberwell, Victoria, Australia
- GSK Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf